CLINICAL TRIAL: NCT01493765
Title: Virtual Temporal Bone Surgery: Defining and Translating Metrics
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Ohio State University (Other)
Responsible Party: Principal Investigator, Gregory Wiet, Associate Professor of Otolaryngology and Biomedical Informatics, Nationwide Children's Hospital
Other Study IDs: R01DC011321-01A1 (NIH)
Record Dates: First submitted 2011-12-13; First posted 2011-12-16 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Focus: Otologic Surgery Training

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Benchmarking: All resident study subjects will drill virtual temporal bones within the computer based system. The performance data will be used to validate the rating metrics and computer scoring process.
  Interventions: Other: Simulator training with expert scoring

INTERVENTIONS:
Other: Simulator training with expert scoring — Residents will be trained using surgical simulation

SUMMARY:
The goal of this project is to improve the efficiency of training and assessment of technical skill in surgical treatment of otologic disease. Through previous funding, we have developed an intuitive virtual simulation environment to be used as an adjuvant for teaching temporal bone surgery. Using direct-volume visualization techniques with integrated stereoscopic display, haptic (force) feedback, and aural simulation, we have achieved a straightforward, low-cost learning environment ready for translation into a practical training and assessment tool. This application challenges and seeks to shift current practice in clinical training by translating the simulation environment into a vehicle for curriculum development, technical skills assessment, and dissemination. The intent is to provide more accessible, inexpensive, safe, and deliberate practice with objective and continuous quantitative, objective assessment in the early stages of training.

DETAILED DESCRIPTION:
The aims of this research include: 1) definition of standardized metrics for otological surgical techniques, 2) the translation of those standards into objective criteria for use in a computer synthesized surgical environment, and 3) the correlation between expert evaluation and computer automated assessment of resident proficiency.

The interactions will be computer-based and include:

Experts will learn to use the system so that they can evaluate the quality of translation of metrics to the simulation environment.

Evaluations will be in the form of anonymous web-based surveys. Experts serve as a focus group.

Residents will use the simulation environment to perform surgical procedures on virtual specimens. Residents will then evaluate the quality of the simulation environment via anonymous web-based surveys.

Experts will use the simulation environment to evaluate and rate the residents performance.

The computer environment will be used to automatically assess and rate the residents performance.

Expert and computer assessment will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Specific knowledge of otologic surgery.

Exclusion Criteria:

* request not to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Novice otology surgeons
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2013-07; Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Performance on a set of validated metrics for temporal bone surgery. | one year
  A collection of metrics designed to measure technical performance during a mastoidectomy will be validated by expert survey. These metrics will be translated to an automated system within the surgical simulation system. Resident subjects will be asked to perform the surgical procedure (mastoidectomy) within the simulation. Experts will then rate the playback of the performances using the validated metrics. These results will be compared to the automated scoring system. A conclusion will be drawn about the accuracy of the automated process compared to the expert rated process.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - UC Irvine, Irvine, California
  - Stanford, Palo Alto, California
  - Iowa, Iowa City, Iowa
  - Henry Ford, Detroit, Michigan
  - Mississippi, Jackson, Mississippi
  - Albert Einstein, The Bronx, New York
  - Duke, Durham, North Carolina
  - The Ohio State University, Columbus, Ohio
  - UT Southwestern, Dallas, Texas
  - Baylor, Houston, Texas